CLINICAL TRIAL: NCT01177124
Title: Mindfulness-Based Stress Reduction (MBSR) Symptom Cluster Trial for Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cecile Lengacher (Other)
Responsible Party: Sponsor-Investigator, Cecile Lengacher, Principal Investigator, University of South Florida
Organization: University of South Florida (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R01CA131080-01A2 (NIH)
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Survivors; Mindfulness-Based Stress Reduction (MBSR); Symptoms; Immune markers
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MBSR 6 Weeks Program (Experimental)
  Interventions: Behavioral: MBSR 6 Weeks Program
- Usual Care (UC) (No Intervention)

INTERVENTIONS:
Behavioral: MBSR 6 Weeks Program — MBSR is a clinical program that provides systematic training to promote stress reduction by self-regulating arousal to stress. The goal of training is to teach participants to become more aware of their thoughts and feelings, and through meditation practice, to have the ability to step back from thoughts and feelings during stressful situations that contribute to increased emotional distress. The intervention incorporates simple yoga, sitting meditation, body scan, and walking meditation in a 6-week program (Kabat-Zinn et al. 1985; Teasdale et al. 1995).
  Other Names: MBSR
  Arms: MBSR 6 Weeks Program

SUMMARY:
The purpose of this study among breast cancer survivors is three-fold: (i) to evaluate the efficacy of the MBSR(BC) program in improving psychological and physical symptoms, quality of life and measures of immune function and a stress hormone (cortisol); (ii) to test whether positive effects achieved from the MBSR(BC) program are mediated through changes in mindfulness and fear of recurrence of breast cancer; and (iii) to evaluate whether positive effects achieved from the MBSR(BC) program are modified by specific patient characteristics measured at baseline.

DETAILED DESCRIPTION:
Breast cancer survivors are living longer and may be living with many symptoms incurred from the disease and its treatment. Survivors from 1 to 2 years off treatment report continued fatigue, depression, pain and sleep disturbances (Kenefick 2006; Byar et al. 2006). Patients often present with several concurrent symptoms (Dodd et al. 2001; Esper and Heidrich 2005). It is believed that symptoms tend to cluster together (two or more concurrent symptoms related to one another and independent of other symptoms) and may have natural associations, similar shared pathways and underlying mechanisms (Barsevick 2007). Currently, little is known about how symptoms cluster in breast cancer survivors after treatment, underlying mechanisms, and if interventions can influence multiple symptoms simultaneously (Lee et al. 2004; Cleeland et al. 2003). Very few studies have tested interventions during post-treatment survivorship (Cimprich et al. 2005; Mishel et al. 2005; Stanton et al. 2005; Scheier et al. 2005). Mindfulness-Based Stress Reduction (MBSR), a standardized form of meditation and yoga, has been shown to be effective in reducing anxiety, depression and stress in patients with chronic pain (Kabat-Zinn et al. 1992; Miller et al. 1995; Teasdale et al. 2000; Kabat-Zinn et al. 1985). Preliminary results from 2 pilot studies conducted by our research team provide support that MBSR for breast cancer survivors may be effective in markedly reducing symptoms, increasing quality of life, and decreasing fears of recurrence (Lengacher et al. 2009; Lengacher et al. 2006). This proposed study builds on our preliminary data of the MBSR Breast Cancer Program (BC) to reduce stress, biological markers of the stress response (pro-inflammatory cytokines) and improve physical, and psychological symptoms and quality of life in breast cancer survivors.

We aim to determine: (i) the extent to which the MBSR(BC) program is efficacious in improving outcomes; (ii) whether positive effects from MBSR(BC) are mediated through increased mindfulness and reduced fear of recurrence; and (iii) if a subgroup of patients can be determined to derive the most benefit from MBSR(BC). Formal specific aims are as follows:

Aim (1). Evaluate the efficacy of the MBSR(BC) program in improving psychological and physical symptoms, quality of life and measures of immune function and a stress hormone (cortisol). We hypothesize that compared to the usual care regimen, patients randomly assigned to the MBSR(BC) program will experience greater improvements at 6 weeks and sustained improvements at 12 weeks in the following:

1. Individual psychological symptoms, including depression anxiety, and perceived stress;
2. Individual physical symptoms, including pain, fatigue and sleep dysfunction;
3. Quality of life;
4. Biological stress markers (pro-inflammatory immune cytokines, cellular adhesion molecules, lymphocyte subsets) and a stress-related hormone (cortisol).

Aim (2). Test whether positive effects achieved from the MBSR(BC) program (defined in 1a-1d) are mediated through changes in mindfulness and fear of recurrence of breast cancer. We hypothesize that:

1. Patients in the MBSR(BC) program will report greater increases in mindfulness and larger reductions in fear of recurrence compared to patients assigned to the usual care regimen.
2. Increased mindfulness will relate directly to improvements in psychological and physical symptoms, quality of life and measures of immune function and a stress hormone (cortisol).
3. Reductions in fear of recurrence will be associated with improvements in psychological and physical symptoms, quality of life and measures of immune function and a stress hormone (cortisol).
4. A primary pathway through which MBSR exerts its positive effects (defined in 1a-1d) will be through increased mindfulness leading to reduced fear of recurrence of cancer.

Aim (3). Evaluate whether positive effects achieved from the MBSR(BC) program (defined in 1a-1d) are modified by specific patient characteristics measured at baseline. We hypothesize that efficacy of the MBSR(BC) program will be greatest among patients with:

1. High anxiety, high perceived stress, low optimism and poor quality of life
2. Specific symptom profiles (i.e. highly distressed patients), as determined by grouping (clustering) patients according to their presenting symptoms.

To achieve this research goal, we have proposed a 2-group randomized clinical trial among 300 breast cancer survivors who have undergone lumpectomy and/or mastectomy and radiation and/or chemotherapy in the past two years. The MBSR(BC) program will be evaluated against a waitlisted usual care regimen (UC), with patient assessments made at baseline, 6 weeks, and 12 weeks. Patient assessments will provide data on depression, state anxiety, perceived stress, fatigue, pain, sleep, symptom severity, quality of life, mindfulness, fear of recurrence, optimism and social support. Additionally, blood and saliva samples will be collected from participants. Biological stress markers will be measured by blood specimen collection; biological stress markers will include pro-inflammatory and anti-inflammatory cytokines (IL-1β, TNF-α, IL-6, IL-10, IL-1-RA, TNF-RA, IL-8, IFN-gamma), cellular adhesion markers (CD11a, CD54, CD62L, CD45RA, CD45RO) and lymphocyte subsets (CD3, CD19, CD16+56). A stress hormone, cortisol, will be measured by saliva specimen collection. The MBSR(BC) intervention is an adapted 6-week program that follows the curriculum of an 8-week program established by Kabat Zinn and Santorelli. Prior to formal hypothesis testing, the distributions of all explanatory and outcome variables, as well as covariates, will be examined. For outcome variables with skewed distributions, appropriate transformations (e.g. square root, logarithmic, etc.) will be performed to satisfy normality requirements for parametric multivariable linear modeling. This will include choosing the transformation which yields the lowest Anderson-Darling score. In instances in which appropriate transformations cannot be achieved, non-parametric methods will be used.

Results from this study will advance conceptual and clinical knowledge of how a stress-reducing intervention impacts symptoms among breast cancer survivors and in whom it may be most efficacious. Determining stress-related biological effects may be applicable to other stress-reducing intervention studies. This symptom and symptom cluster assessment and intervention model will further our understanding of biology and behavior and test a predictive and personalized model of health care.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older
* Diagnosed with Stage 0, I, II, or III breast cancer
* Undergone lumpectomy and/or mastectomy and are at 2 weeks from end of treatment with adjuvant radiation and/or chemotherapy or are a maximum of 2 years out from completion of such treatment
* Ability to read and speak English at the 8th grade level or above to respond to survey questions

Exclusion Criteria:

* Advanced stage (IV) cancer
* Current psychiatric diagnosis
* Recurrent treatment for prior breast cancer

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-02; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of the MBSR(BC) program in improving psychological and physical symptoms, quality of life and measures of immune function and a stress hormone (cortisol) | Baseline, 6 weeks and 12 weeks

SECONDARY OUTCOMES:
To test whether positive effects achieved from the MBSR(BC) program are mediated through changes in mindfulness and fear of recurrence of breast cancer | Baseline, 6 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cecile A Lengacher, RN, PhD, Principal Investigator — University of South Florida
Locations (3):
- United States (3):
  - Carol and Frank Morsani Center for Advanced Healthcare, Tampa, Florida
  - Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of South Florida, Tampa, Florida

REFERENCES:
- [Background] Kenefick AL. Patterns of symptom distress in older women after surgical treatment for breast cancer. Oncol Nurs Forum. 2006 Nov 3;33(2):327-35. doi: 10.1188/06.ONF.327-335. PMID 16518448
- [Background] Byar KL, Berger AM, Bakken SL, Cetak MA. Impact of adjuvant breast cancer chemotherapy on fatigue, other symptoms, and quality of life. Oncol Nurs Forum. 2006 Jan 1;33(1):E18-26. doi: 10.1188/06.ONF.E18-E26. PMID 16470230
- [Background] Dodd MJ, Miaskowski C, Paul SM. Symptom clusters and their effect on the functional status of patients with cancer. Oncol Nurs Forum. 2001 Apr;28(3):465-70. PMID 11338755
- [Background] Esper P, Heidrich D. Symptom clusters in advanced illness. Semin Oncol Nurs. 2005 Feb;21(1):20-8. doi: 10.1053/j.soncn.2004.10.004. PMID 15807053
- [Background] Barsevick AM. The elusive concept of the symptom cluster. Oncol Nurs Forum. 2007 Sep;34(5):971-80. doi: 10.1188/07.ONF.971-980. PMID 17878126
- [Background] Lee BN, Dantzer R, Langley KE, Bennett GJ, Dougherty PM, Dunn AJ, Meyers CA, Miller AH, Payne R, Reuben JM, Wang XS, Cleeland CS. A cytokine-based neuroimmunologic mechanism of cancer-related symptoms. Neuroimmunomodulation. 2004;11(5):279-92. doi: 10.1159/000079408. PMID 15316238
- [Background] Cleeland CS, Bennett GJ, Dantzer R, Dougherty PM, Dunn AJ, Meyers CA, Miller AH, Payne R, Reuben JM, Wang XS, Lee BN. Are the symptoms of cancer and cancer treatment due to a shared biologic mechanism? A cytokine-immunologic model of cancer symptoms. Cancer. 2003 Jun 1;97(11):2919-25. doi: 10.1002/cncr.11382. PMID 12767108
- [Background] Cimprich B, Janz NK, Northouse L, Wren PA, Given B, Given CW. Taking CHARGE: A self-management program for women following breast cancer treatment. Psychooncology. 2005 Sep;14(9):704-17. doi: 10.1002/pon.891. PMID 15651055
- [Background] Mishel MH, Germino BB, Gil KM, Belyea M, Laney IC, Stewart J, Porter L, Clayton M. Benefits from an uncertainty management intervention for African-American and Caucasian older long-term breast cancer survivors. Psychooncology. 2005 Nov;14(11):962-78. doi: 10.1002/pon.909. PMID 15712339
- [Background] Stanton AL, Ganz PA, Kwan L, Meyerowitz BE, Bower JE, Krupnick JL, Rowland JH, Leedham B, Belin TR. Outcomes from the Moving Beyond Cancer psychoeducational, randomized, controlled trial with breast cancer patients. J Clin Oncol. 2005 Sep 1;23(25):6009-18. doi: 10.1200/JCO.2005.09.101. PMID 16135469
- [Background] Scheier MF, Helgeson VS, Schulz R, Colvin S, Berga S, Bridges MW, Knapp J, Gerszten K, Pappert WS. Interventions to enhance physical and psychological functioning among younger women who are ending nonhormonal adjuvant treatment for early-stage breast cancer. J Clin Oncol. 2005 Jul 1;23(19):4298-311. doi: 10.1200/JCO.2005.05.362. PMID 15994143
- [Background] Kabat-Zinn J, Massion AO, Kristeller J, Peterson LG, Fletcher KE, Pbert L, Lenderking WR, Santorelli SF. Effectiveness of a meditation-based stress reduction program in the treatment of anxiety disorders. Am J Psychiatry. 1992 Jul;149(7):936-43. doi: 10.1176/ajp.149.7.936. PMID 1609875
- [Background] Miller JJ, Fletcher K, Kabat-Zinn J. Three-year follow-up and clinical implications of a mindfulness meditation-based stress reduction intervention in the treatment of anxiety disorders. Gen Hosp Psychiatry. 1995 May;17(3):192-200. doi: 10.1016/0163-8343(95)00025-m. PMID 7649463
- [Background] Teasdale JD, Segal ZV, Williams JM, Ridgeway VA, Soulsby JM, Lau MA. Prevention of relapse/recurrence in major depression by mindfulness-based cognitive therapy. J Consult Clin Psychol. 2000 Aug;68(4):615-23. doi: 10.1037//0022-006x.68.4.615. PMID 10965637
- [Background] Kabat-Zinn J, Lipworth L, Burney R. The clinical use of mindfulness meditation for the self-regulation of chronic pain. J Behav Med. 1985 Jun;8(2):163-90. doi: 10.1007/BF00845519. PMID 3897551
- [Background] Lengacher CA, Johnson-Mallard V, Post-White J, Moscoso MS, Jacobsen PB, Klein TW, Widen RH, Fitzgerald SG, Shelton MM, Barta M, Goodman M, Cox CE, Kip KE. Randomized controlled trial of mindfulness-based stress reduction (MBSR) for survivors of breast cancer. Psychooncology. 2009 Dec;18(12):1261-72. doi: 10.1002/pon.1529. PMID 19235193
- [Background] Lengacher C, Gaurkee D, Mierzejewski A, et al. Feasibility of MBSR in early stage breast cancer recovery, a pilot study. Breast Cancer Research and Treatment. 2006;100(1):s289-290.
- [Background] Teasdale JD, Segal Z, Williams JM. How does cognitive therapy prevent depressive relapse and why should attentional control (mindfulness) training help? Behav Res Ther. 1995 Jan;33(1):25-39. doi: 10.1016/0005-7967(94)e0011-7. PMID 7872934
- [Derived] Lengacher CA, Gruss LF, Kip KE, Reich RR, Chauca KG, Moscoso MS, Joshi A, Tinsley S, Shani B, Cousin L, Khan CP, Goodman M, Park JY. Mindfulness-based stress reduction for breast cancer survivors (MBSR(BC)): evaluating mediators of psychological and physical outcomes in a large randomized controlled trial. J Behav Med. 2021 Oct;44(5):591-604. doi: 10.1007/s10865-021-00214-0. Epub 2021 May 7. PMID 33963420
- [Derived] Reich RR, Lengacher CA, Alinat CB, Kip KE, Paterson C, Ramesar S, Han HS, Ismail-Khan R, Johnson-Mallard V, Moscoso M, Budhrani-Shani P, Shivers S, Cox CE, Goodman M, Park J. Mindfulness-Based Stress Reduction in Post-treatment Breast Cancer Patients: Immediate and Sustained Effects Across Multiple Symptom Clusters. J Pain Symptom Manage. 2017 Jan;53(1):85-95. doi: 10.1016/j.jpainsymman.2016.08.005. Epub 2016 Oct 5. PMID 27720794
- [Derived] Lengacher CA, Reich RR, Paterson CL, Ramesar S, Park JY, Alinat C, Johnson-Mallard V, Moscoso M, Budhrani-Shani P, Miladinovic B, Jacobsen PB, Cox CE, Goodman M, Kip KE. Examination of Broad Symptom Improvement Resulting From Mindfulness-Based Stress Reduction in Breast Cancer Survivors: A Randomized Controlled Trial. J Clin Oncol. 2016 Aug 20;34(24):2827-34. doi: 10.1200/JCO.2015.65.7874. Epub 2016 May 31. PMID 27247219
- [Derived] Lengacher CA, Reich RR, Paterson CL, Jim HS, Ramesar S, Alinat CB, Budhrani PH, Farias JR, Shelton MM, Moscoso MS, Park JY, Kip KE. The effects of mindfulness-based stress reduction on objective and subjective sleep parameters in women with breast cancer: a randomized controlled trial. Psychooncology. 2015 Apr;24(4):424-32. doi: 10.1002/pon.3603. Epub 2014 Jun 18. PMID 24943918